CLINICAL TRIAL: NCT00000578
Title: NHLBI/NICHD Collaborative Studies of Asthma in Pregnancy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Treatment
Other Study IDs: 216
Record Dates: First submitted 1999-10-27; First posted 1999-10-28 (Estimated); Last update posted 2016-07-12 (Estimated); Status verified 2005-02

CONDITIONS: Asthma; Lung Diseases
MeSH Terms: conditions — Asthma; Lung Diseases | interventions — Theophylline; Beclomethasone

INTERVENTIONS:
Drug: theophylline
Drug: beclomethasone

SUMMARY:
To conduct a collaborative program of research on asthma and pregnancy consisting of two studies: the Asthma in Pregnancy Study (APS) was an observational study to evaluate relationships between asthma severity and treatment programs and perinatal outcome, and the Asthma Therapy in Pregnancy Trial (ATPT) was a randomized clinical trial of inhaled beclomethasone versus theophylline in the treatment of moderate asthma during pregnancy. Both studies were conducted in the Maternal-Fetal Medicine Unit (MFMU) Network, an ongoing group of participating obstetric centers supported by the National Institute of Child Health and Human Development. Studies were co-funded by the NHLBI.

DETAILED DESCRIPTION:
BACKGROUND:

Asthma is one of the most common illnesses that complicates pregnancy. Asthma complicates at least 4 percent of all pregnancies; however, because at least 10 percent of the population appears to have nonspecific airway hyper-responsiveness, the true prevalence may be much higher.

Asthma can produce serious maternal and fetal complications. A number of investigators have reported an increased incidence of pre-eclampsia, gestational hypertension, hyperemesis gravidarum, vaginal hemorrhage, toxemia, and induced and complicated labor. Fetal complications include increased risk of perinatal mortality, prematurity, low birth weight, and neonatal hypoxia. In contrast, several studies have failed to confirm some or all of these previous observations. Patients with severe asthma may have the greatest risk for complications during pregnancy, in addition to the risk of maternal morbidity from the asthma. For example, it has been shown that reduced pulmonary function in asthmatic women is associated with an increased likelihood of intrauterine growth retardation. On the other hand, studies in which asthma was successfully controlled have resulted in pregnancy outcomes similar to the general population.

The mechanisms by which asthma may have adverse perinatal effects are not well known. Poor control of asthma leading to chronic or episodic fetal hypoxia is thought to be important. Medications used in asthma treatment may also play a role, although the limited data suggests minimal or no effects. In addition, it is possible that extrapulmonary autonomic nervous system abnormalities, such as uterine muscle hyperreactivity, could contribute to pre-term delivery or gestational hypertension independent of asthma control or therapy.

Unfortunately, previous studies have been limited by relatively small numbers. Few studies have controlled for factors known to affect infant birth weight, such as maternal race, height, weight, parity, nutrition, and cigarette smoking. Particularly, race may be an important contributing factor in assessing the relationship between asthma and pregnancy outcomes, since Blacks of both sexes are twice as likely to be hospitalized from asthma and three times as likely to die from asthma as whites.

Under the auspices of the National Asthma Education Program (NAEP), a Working Group on Asthma and Pregnancy developed a statement regarding the treatment of asthma during pregnancy. In its deliberations, the Working Group noted the paucity of data on the relative contributions of biological, social, and environmental factors on asthma in pregnant women, as well as the lack of data on the efficacy and safety of commonly used asthma therapies in pregnancy.

DESIGN NARRATIVE:

The Asthma in Pregnancy Study evaluated the relationship between maternal asthma severity and control. The primary objective was to determine the frequency of preterm delivery <32 weeks among moderate and severe asthmatics compared to non-asthmatic controls. The incidence of small-for-gestational-age infants in women with mild and moderate asthma was a secondary outcome. Other independent variables included type of medications used, race, socioeconomic status, height, weight, parity, nutrition, smoking, other substance abuse, and prenatal care. Secondary outcomes included birth weight and prematurity, maternal pre-eclampsia, gestational hypertension, and asthma morbidity. The study began February 1,1995 and patient recruitment continued for 46 months or less.

The Asthma Therapy in Pregnancy Trial was a randomized, double-blind, controlled clinical trial which began recruitment in November, 1996, with enrollment lasting 44 months. Patients were randomized to receive either active oral theophylline and a placebo beclomethasone inhaler or an active beclomethasone inhaler and placebo oral theophylline. Albuterol was used for relief of symptoms. The primary outcome measure was incidence of Emergency Department visits or hospitalizations during pregnancy. Secondary outcome measures included birth weight, incidence of small-for-gestational-age infants, gestational hypertension, pre-eclampsia, lung function, daily peak flow, and quality of life. Patients were seen monthly for measurements of fetal growth, morbidity, and lung function. Extensive interviews were conducted with each patient at the first prenatal visit, in the third trimester, and shortly before birth.

The study completion date listed in this record was obtained from the "Completed Date" entered in the Query View Report System (QVR).

ELIGIBILITY:
Asthmatic pregnant women.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Dates: Start 1994-04; Study Completion 2000-10 (Actual)

REFERENCES:
- [Background] Wright LL, McNellis D. National Institute of Child Health and Human Development (NICHD)-sponsored Perinatal Research Networks. Semin Perinatol. 1995 Apr;19(2):112-23. doi: 10.1016/s0146-0005(05)80031-x. No abstract available. PMID 7604302
- [Background] Dombrowski MP, Schatz M, Wise R, Momirova V, Landon M, Mabie W, Newman RB, McNellis D, Hauth JC, Lindheimer M, Caritis SN, Leveno KJ, Meis P, Miodovnik M, Wapner RJ, Paul RH, Varner MW, O'Sullivan MJ, Thurnau GR, Conway DL; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network and the National Heart, Lung, and Blood Institute. Asthma during pregnancy. Obstet Gynecol. 2004 Jan;103(1):5-12. doi: 10.1097/01.AOG.0000103994.75162.16. PMID 14704237
- [Background] Dombrowski MP, Schatz M, Wise R, Thom EA, Landon M, Mabie W, Newman RB, McNellis D, Hauth JC, Lindheimer M, Caritis SN, Leveno KJ, Meis P, Miodovnik M, Wapner RJ, Varner MW, O'Sullivan MJ, Conway DL; National Institute of Child Health and Human Development Maternal-Fetal Medicine Units Network; National Heart, Lung, and Blood Institute. Randomized trial of inhaled beclomethasone dipropionate versus theophylline for moderate asthma during pregnancy. Am J Obstet Gynecol. 2004 Mar;190(3):737-44. doi: 10.1016/j.ajog.2003.09.071. PMID 15042007